CLINICAL TRIAL: NCT06079801
Title: Bilateral DLPC tDCS: a New Potential Neuromodulatory Strategy in Drug-resistant Migraine
Brief Title: Bilateral DLPC tDCS in Drug-resistant Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Intervención en Neurociencias (Other)
Responsible Party: Principal Investigator, Michele Dileone, MD, PhD, Principal Investigator, Neurologist, Clínica de Intervención en Neurociencias
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ClinicaIN01
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Migraine
Keywords: migraine; drug-resistant; tDCS; DLPC; Neuromodulation; anti CGRP
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Real tDCS (Experimental): Patients will undergo real tDCS applied to both DLPC. Two daily sessions of 20 minutes each were administered (40 minutes a day in total), with a 5-minutes break in between, 5 days a week (Monday to Friday) and with 20 tDCS sessions in total for participant
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham tDCS (Placebo Comparator): Patients will undergo sham tDCS applied to both DLPC. Two daily sessions of 20 minutes each were administered (40 minutes a day in total), with a 5-minutes break in between, 5 days a week (Monday to Friday) and with 20 tDCS sessions in total for participant
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- anti-CGRP (Active Comparator): Patients will undergo anti-CGRP treatment
  Interventions: Drug: anti-CGRP-mAbs

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — TDCS was delivered by a DC-Stimulator (Newronika, Italy) over both DLPC. The electrodes (35 cm2) were soaked in 0.9% NaCl. The anode was positioned on the left dorsolateral prefrontal cortex and the cathode on the right dorsolateral prefrontal cortex.
  Arms: Real tDCS; Sham tDCS
Drug: anti-CGRP-mAbs — CGRP-mAbs have been the first target-driven treatment to be approved for migraine prevention. Their efficacy and safety have been demonstrated in randomized controlled trials (RCT) as well as, in real-world evidence (RWE) studies
  Arms: anti-CGRP

SUMMARY:
The goal of this clinical trial is to study and describe the effects of bilateral tDCS applied to dorso-lateral-prefrontal cortex (DLPC) in patients with drug-resistant migraine in terms of reduction in frequency of pain, impact of pain in daily life, quality of sleep and psychological measures. We finally planned to include high frequency and chronic migraine patients.

The main questions it aims to answer are:

* Will bilateral DLPC tDCS be feasible, well tolerated and safe in drug resistant migraine patients?
* Will bilateral DLPC tDCS be effective in reducing pain frequency, intensity and its impact in daily life activities?
* Will bilateral DLPC tDCS be effective in ameliorating sleep and psychological associated symptoms?
* Will bilateral DLPC tDCS be such effective in reducing pain frequency, intensity and its impact in daily life activities as anti-CGRP treatments?

Participants will undergo 2 tDCS sessions daily for 2 consecutive weeks. Patients will be blinded to treatment and will be divided in two groups (real vs placebo). A third group of patients, age-matched to the other two, will undergo anti-CGRP treatment. Patients will be asked to complete Patient-Reported Outcomes (PROMs) scales at baseline, one week after the end of the treatment and at 6 months after the end of the treatment.

Researchers (blinded to the treatment) will compare the group that underwent real tDCS treatment vs the one that underwent placebo tDCS vs the one that underwent anti-CGRP drugs to see if bilateral DLPC tDCS is effective in reducing migraine frequency, intensity and impact and if bilateral DLPC tDCS is such effective as anti-CGRP treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of high-frequency and/or chronic migraines, according to the diagnostic criteria of the ICHD-III,
* failure to more than 3 preventive drugs
* stable pharmacological treatment (> 6 months without changes),
* absence of other neurological or medical pathological conditions,
* written informed consent.

Exclusion Criteria:

* seizures
* significant cognitive impairment that prevents following orders and understanding instructions (Mini-Mental State Examination < 23)
* pregnancy
* aphasia or limitations in communication,
* metallic cranial implants
* another neurological or psychiatric pathology
* diagnosis of another type of migraine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Migraine attacks monthly frequency | baseline, 2 weeks after the end of the treatment, 6 months
  Patients will report migraine monthly frequency for the 3 different time-points
Headache Impact Test (HIT-6) score | baseline, 2 weeks after the end of the treatment, 6 months
  HIT-6 is a tool used to measure the impact headaches have on patient's ability to function on the job, at school, at home and in social situations.
Pain killer drugs monthly taken | baseline, 2 weeks after the end of the treatment, 6 months
  Patients will report pain-killer drugs taken during a month for the 3 different time-points

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | baseline, 2 weeks after the end of the treatment, 6 months
  PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.
Brief Symptom Inventory (BSI) | baseline, 2 weeks after the end of the treatment, 6 months
  The Brief Symptom Inventory (BSI) consists of 53 items covering nine symptom dimensions: Somatization, Obsession-Compulsion, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation and Psychoticism; and three global indices of distress: Global Severity Index, Positive Symptom Distress Index, and Positive Symptom Total. The global indices measure current or past level of symptomatology, intensity of symptoms, and number of reported symptoms, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica de Intervencion en Neurociencias, Talavera de la Reina, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No
We will publish results of the study and we will provide more information for reviewers if required